CLINICAL TRIAL: NCT00552864
Title: High Thoracic Epidural Anesthesia and Postoperative Analgesia With Ropivacaine or Levobupivacaine for Coronary Surgery: A Prospective Randomized Double-Blind Comparison
Brief Title: Comparison of Ropivacaine and Levobupivacaine in High Thoracic Epidural Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCMAneste001
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Coronary Artery Bypass; Epidural Anesthesia
MeSH Terms: interventions — Ropivacaine; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- R (Active Comparator)
  Interventions: Drug: Ropivacaine
- L (Active Comparator)
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Ropivacaine — 0.5% epidural bolus injection (0.1 mL kg-1) with sufentanil 2.5 µg mL-1 before general anesthesia induction, followed by 0.2% infusion (0.1 mL kg-1 h-1) with sufentanil 1 µg mL-1 throughout surgery; in ICU, 0.1% epidural infusion with sufentanil 1µg mL-1 at 0.1 mL kg-1 h-1 and the rate is modified following this protocol: on awakening (Ramsay 2) VAS on coughing is evaluated: if it is 4 the infusion rate is not changed, if the VAS is ≥ 4 the rate is increased by 2 mL h-1 after giving a 2 mL bolus and VAS is checked again 30 minutes later, if it is ≤ 4 the infusion rate is decreased by 2 mL h-1.
  Other Names: Naropina
  Arms: R
Drug: Levobupivacaine — 0.5% epidural bolus injection (0.1 mL kg-1) with sufentanil 2.5 µg mL-1 before general anesthesia induction, followed by 0.2% infusion (0.1 mL kg-1 h-1) with sufentanil 1 µg mL-1 throughout surgery; in ICU, 0.1% epidural infusion with sufentanil 1µg mL-1 at 0.1 mL kg-1 h-1 and the rate is modified following this protocol: on awakening (Ramsay 2) VAS on coughing is evaluated: if it is 4 the infusion rate is not changed, if the VAS is ≥ 4 the rate is increased by 2 mL h-1 after giving a 2 mL bolus and VAS is checked again 30 minutes later, if it is ≤ 4 the infusion rate is decreased by 2 mL h-1.
  Other Names: Chirocaina
  Arms: L

SUMMARY:
In High Thoracic Epidural Anesthesia (HTEA) the use of a local anesthetic (LA) with low cardiac toxicity is crucial as myocardial contractility is often already seriously impaired. The aim of this study is to compare the efficacy, doses and side effects of ropivacaine and levobupivacaine in patients submitted to coronary artery bypass graft with HTEA and general anesthesia. The primary end point is the amount of LA drug required to maintain a VAS < 4 when coughing in the first 24 postoperative hours.

DETAILED DESCRIPTION:
The use of high thoracic epidural, combined with general anesthesia (HTEA) in patients undergoing cardiac surgery has become increasing popular in recent years. In fact, this technique is potentially beneficial because of the attenuation of the stress response to surgery, the sympathetic tone reduction and the excellent postoperative analgesia.Patients submitted to coronary artery bypass graft will be randomly allocated to receive high epidural block with ropivacaine (R) or levobupivacaine (L), supplemented with sufentanil, during and after surgery. Postoperatively, the rate of epidural infusion will be modified to maintain a VAS score less than 4 in the thoracic area when coughing. VAS, total amount and rate of epidural drug infusion, MAP, total amount and rate of norepinephrine infusion and motor block will be recorded on arrival in the ICU, on awakening and after 4, 8, 12, 24 hours. Additionally, the onset time of the epidural sensory block, the time of awakening and the time on ventilator will be recorded as well as episodes of postoperative nausea and vomiting (PONV) and pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for coronary artery bypass grafting
* with stable angina
* left ventricular ejection fraction > 30%
* age > 18 years
* having signed a written informed consent.
* Prothrombin Time (PT) > 80% and Partial Thromboplastin Time (PTT) within the normal range, and platelet counts (PLT) > 100.000 /mL

Exclusion Criteria:

* emergency operation
* known coagulation disorders or recent thrombolytic therapy
* angina on arrival in the operating room
* acute myocardial infarction within the previous seven days
* clinically significant associated valvular disease
* known neuraxial pathology
* patients participating in other clinical research protocols.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2003-01; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
The amount of local anesthetic drug (mg) required to maintain a visual analog scale score for pain (VAS) < 4 when coughing. | the first 24 postoperative hours

SECONDARY OUTCOMES:
- The onset time of a T1-T6 block after the bolus. - the amount of norepinephrine needed to maintain MAP > 70. - differences in motor block. - side effects. | The first 24 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: Luca Salvi, MD, Principal Investigator — Department of Anesthesia & ICU. IRCCS Centro Cardiologico Monzino.
Locations (1):
- Department of Anesthesia & ICU. IRCCS Centro Cardiologico Monzino, Milan, Italy

REFERENCES:
- [Background] Olivier JF, Le N, Choiniere JL, Prieto I, Basile F, Hemmerling T. Comparison of three different epidural solutions in off-pump cardiac surgery: pilot study. Br J Anaesth. 2005 Nov;95(5):685-91. doi: 10.1093/bja/aei238. Epub 2005 Sep 23. PMID 16183682
- [Background] Casati A, Putzu M. Bupivacaine, levobupivacaine and ropivacaine: are they clinically different? Best Pract Res Clin Anaesthesiol. 2005 Jun;19(2):247-68. doi: 10.1016/j.bpa.2004.12.003. PMID 15966496